CLINICAL TRIAL: NCT01698996
Title: A Randomized Blinded Trial of Abscess Management With Packing vs No Packing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Amit Shah, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102928
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Uncomplicated Cutaneous Abscess
Keywords: abscess; packing; emergency medicine; wound care; incision and drainage
MeSH Terms: conditions — Abscess; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Packing (Active Comparator): No Packing
  Interventions: Procedure: Packing vs No Packing
- Packing (Experimental): Packing
  Interventions: Procedure: Packing vs No Packing

INTERVENTIONS:
Procedure: Packing vs No Packing

SUMMARY:
Adult patients presenting to the emergency department with superficial cutaneous abscesses will be randomized after incision and drainage to standard care with wound packing or no packing to determine if there is a difference in the proportion of complications between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Abscess ≤ 5cm in diameter
* Truncal or extremity location

Exclusion Criteria:

* Post-operative abscess (abscess in location of operative incision, operation within the last 4 months)
* HIV/immunocompromised/transplant recipient/chronic oral steroid use
* Fever at triage (temp ≥38 degrees Celsius)
* Abscess secondary to Crohn's
* Multiple abscesses requiring drainage
* Prior participation in the study for the same abscess
* Incision and drainage performed with no packing required, or where abscess cavity is <1 cm max diameter
* Bartholins/perigenital, perianal, or facial abscesses
* Complicated abscesses (fistula, suspicion of muscular extension, consultation/direct referral to general surgery)
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of complications (defined as a composite of the following: need for repeat incision and drainage by physician, need for admission to hospital, or need for escalation to intravenous antibiotics) | 7 days

SECONDARY OUTCOMES:
Proportion of wounds "closed" at 1 week (wound size <0.5 cm length and depth and no drainage) | 7 days

OTHER OUTCOMES:
Proportion of wounds "closed" at 2 weeks (wound size <0.5 cm length and depth and no drainage) | 14 days
Pain scores (daily pain scores for first week from patient diary) | 7 days
Amount of Pain Medication Used | 7 days
Resources Utilized | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Amit P Shah, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada